CLINICAL TRIAL: NCT05704582
Title: A Randomized Controlled Trial Comparing Avatar Intervention to an Addiction Supportive Intervention to Reduce Cannabis Use in Patients With Psychotic Disorders
Brief Title: RCT Comparing Avatar Intervention to Supportive Intervention to Reduce Cannabis Use in Patients With Psychotic Disorders
Acronym: AC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MP-12-2023-3234
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorders; Cannabis Use Disorder; Mental Health Disorder
Keywords: cannabis; virtual reality intervention; psychotic disorders; substance use disorders
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders; Marijuana Abuse; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar Intervention (Experimental): The Avatar Intervention will take place over 8 consecutive weeks, with one session per week. Additional sessions (up to a maximum of 4 sessions) will be offered if needed. Each session will last approximately 60 minutes. The goal of the intervention will be to help you reduce cravings related to your cannabis use with the use of virtual reality and avatars.
  Interventions: Other: Avatar Intervention
- Addiction supportive intervention (Active Comparator): The Addiction supportive intervention will take place over 8 consecutive weeks, with one session per week. Additional sessions (up to a maximum of 4 sessions) will be offered if needed. Each session will last approximately 60 minutes. The goal of the intervention will be to help you reduce cravings related to your cannabis use.
  Interventions: Other: Addiction supportive intervention

INTERVENTIONS:
Other: Avatar Intervention — 8 weekly sessions of 60 minutes. Possibility of 4 additional sessions.
  Other Names: Avatar-CUD
  Arms: Avatar Intervention
Other: Addiction supportive intervention — 8 weekly sessions of 60 minutes. Possibility of 4 additional sessions.
  Arms: Addiction supportive intervention

SUMMARY:
The goal of this clinical trial is to conduct a single-blind randomized controlled trial to verify whether the Avatar Intervention has greater efficacy over supportive intervention to reduce cannabis use in patients with psychotic disorders.

DETAILED DESCRIPTION:
Psychotic disorders (PD) are characterized by a loss of contact with reality. Cannabis use is one of the key factors leading to psychiatric re-hospitalization in PD. In these populations, cannabis use is also associated with depressive symptoms, medication non-compliance, hostility as well as reduced quality of life. Unfortunately, there is no evidence-based intervention available for the treatment of cannabis use disorder (CUD) in this population. Novel interventions for CUD are thus critically needed. Virtual reality-based therapies are a promising avenue that allow patients to try novel strategies in real time instead of having to learn abstract rules. To fill a clinical need, the investigators have created a distinctive intervention for CUD in patients with PD. The Avatar Intervention displays strong experiential and relational components that are crucially missing in conventional interventions.

Hence, the primary outcomes are reductions in cannabis use, cannabis use disorder severity, and increased quality of life. The investigators will also explore whether the greater improvements attributable to the Avatar Intervention persist in time, and perform analyses on sex/gender, motivation to change cannabis habits, psychotic relapses, and THC metabolite levels.

Noteworthily, cannabis-related hospitalizations have been identified as one of the core indicators to measure the success of cannabis legalization. As a result, there is a pressing need to design innovative interventions that could have a significant impact on this costly and prime outcome. As there is no evidence-based therapeutic options for CUD in patients with PD, the current trial will contribute to the validation of a novel approach and create new therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Males or females over 18 years of age who meet the DSM-5 criteria for CUD (≥4 criteria) ;
* Patients will meet the DSM-5 criteria for schizophrenia, schizoaffective disorder, or bipolar disorder with psychotic symptoms. Diagnoses will be established with the Structured Interview for DSM-5 (SCID-5).

Exclusion Criteria:

* Current SUD for a substance other than cannabis ;
* Ongoing pharmacological or psychological treatment for CUD ;
* Ongoing detoxification for cannabis withdrawal ;
* Presence of neurological disorders ;
* Presence of a severe and unstable physical illness ;
* Inability to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use (Timeline Follow-Back) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  A standardized tool consisting of asking the patients how many joints they smoked each day of the week during the past week.

SECONDARY OUTCOMES:
Change in the severity of the cannabis use disorder (Cannabis Use Problems Identification Test - CUPIT) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  16-item self-reported questionnaire assessing cannabis use and dependence; Range 3-82, higher values indicating a more severe cannabis use disorder
Change in quality of life(Quality of Life Enjoyment and Satisfaction Questionnaire - QLESQ-SF & Quality of Life Scale - QLS) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  QLESQ-SF: 16-item self-reported scale measuring enjoyment and satisfaction experienced during the past week in various areas of daily functioning; Range 14-70, Higher values indicate a better satisfaction of life
  QLS: 21-item scale based on a semistructured interview designed to assess deficit symptoms; Range 0-126, higher values indicate a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, MD, PhD, Principal Investigator — University of Montreal, Institut universitaire en santé mentale de Montréal; Stephane Potvin, PhD, Principal Investigator — University of Montreal, Institut universitaire en santé mentale de Montréal; Emmanuel Stip, MD, MSc, Study Chair — United Arab Emirates University; Amal Abdel Baki, MD, MSc, Study Chair — University of Montreal, Centre hospitalier de l'Université de Montréal; Robert-Paul Juster, PhD, Study Chair — University of Montreal, Institut universitaire en santé mentale de Montréal; Marie-Hélène Goulet, PhD, Study Chair — University of Montreal, Institut universitaire en santé mentale de Montréal; Luigi De Benedictis, MD, Study Chair — Institut universitaire en santé mentale de Montréal
Locations (1):
- Research center of the Institut universitaire en santé mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No